CLINICAL TRIAL: NCT00072124
Title: A Prospective Random Assignment Trial Comparing Complete Metastasectomy to Chemotherapy for Selected Patients With Stage IV Melanoma
Brief Title: Dacarbazine and/or Cisplatin Compared With Complete Metastasectomy in Treating Patients With Stage IV Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000335471; NCI-03-C-0279; NCT00068939 (obsolete NCT alias)
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2005-01

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Cisplatin; Dacarbazine

INTERVENTIONS:
Drug: cisplatin
Drug: dacarbazine
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as dacarbazine and cisplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Complete metastasectomy may be an effective treatment for metastatic melanoma and may improve quality of life and help patients live longer and more comfortably. It is not yet known whether complete metastasectomy is more effective than chemotherapy in treating stage IV melanoma.

PURPOSE: This randomized phase III trial is studying dacarbazine and/or cisplatin to see how well they work compared to complete metastasectomy in treating patients with stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare overall survival in patients with stage IV melanoma treated with complete metastasectomy vs dacarbazine and/or cisplatin.

Secondary

* Compare time to progression in patients treated with these regimens.
* Determine the response rate in patients treated with dacarbazine and/or cisplatin.
* Compare the morbidity and quality of life of patients treated with these regimens.

OUTLINE: This is a randomized study. Patients are stratified according to prior exposure to dacarbazine and cisplatin (yes vs no) and number of sites of metastases (1 vs 2 or more). Patients are randomized to 1 of 2 treatment arms.

* Arm I (surgery): Patients undergo complete metastasectomy. Patients with disease progression after surgery may undergo repeat resection or may receive dacarbazine and/or cisplatin as in arm II.
* Arm II (systemic therapy): Patients receive dacarbazine IV over 30-60 minutes and/or cisplatin IV over 30 minutes on days 1, 2, 3, 22, 23, and 24 (1 course). Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive at least 1 additional course of chemotherapy beyond CR and are eligible for other investigational strategies.

Quality of life is assessed at baseline, at 3 and 6 months, and at 1 year.

Patients are followed every 3-4 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 74 patients (37 per treatment arm) will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic melanoma

  * Solitary pulmonary nodule may not be sole site of metastatic disease
  * No disease limited to subcutaneous, cutaneous, or peripheral nodal (neck, axillary, groin, or iliac nodes) sites only
* Measurable disease
* Disease progression during or after prior interleukin-2 (IL-2)-based therapy OR ineligible for high-dose IL-2 therapy
* Metastatic disease amenable to complete surgical resection

  * Less than 5% estimated mortality from surgery
  * Prior complete metastasectomy allowed provided disease did not recur within 6 months after surgery
* No primary ocular or mucosal melanoma
* No brain metastases

PATIENT CHARACTERISTICS:

Age

* 16 and over

Performance status

* ECOG 0-2

Life expectancy

* More than 3 months

Hematopoietic

* WBC at least 3,000/mm^3 OR
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No coagulation disorder

Hepatic

* Hepatitis B surface antigen negative
* Hepatitis C antibody negative

Renal

* Creatinine no greater than 1.6 mg/dL OR
* Creatinine clearance at least 70 mL/min
* No major medical illness of the renal system

Cardiovascular

* No major medical illness of the cardiovascular system

Pulmonary

* No major medical illness of the respiratory system

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No active systemic infection
* No form of primary or secondary immunodeficiency

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* No concurrent palliative radiotherapy

Surgery

* See Disease Characteristics
* No concurrent palliative surgery

Other

* More than 3 weeks since prior therapy for melanoma (except surgery)
* No other concurrent therapy for melanoma

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-09; Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard M. Sherry, MD, Study Chair — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States